CLINICAL TRIAL: NCT04862546
Title: Effect of Acupuncture Points Laser Versus Tap Water Iontophoresis on Hyperhidrosis
Brief Title: Laser Acupuncture Versus Tap Water Iontophoresis on Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Kadry, Lecture of Physical Therapy, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LaserAcupuncture
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Acupoint (Experimental): Laser will be performed 3 times per week for 2-week measurement. The duration of each cession will be 10 minutes treatment.
  Interventions: Device: Laser Acupoint
- Tap water iontophoresis (Active Comparator): Tap water iontophoresis will be performed 3 times per week for 2-weeks. The duration of each cession will be 20 minutes treatment session.
  Interventions: Device: Tap water iontophoresis

INTERVENTIONS:
Device: Laser Acupoint — Step 1: The subject was in sitting position and exposure area for applying laser then therapist use tap measurement to find the point. Parameters was used in this study : PROBE :ML A1\25 TIME:01:00 FREQUENCY: 10000Hz (25mw), DUTY-CYCLE:100% DENESITY: 1J\CM2 AREA :1CM2 Step 2: Apply laser on acupuncture points by using 10000HZ for 1 minute for every point. Totally cession: 10 minutes Step 3: ensure that all point done Repeat all steps for every subject
  Arms: Laser Acupoint
Device: Tap water iontophoresis — Enough tap water is placed in the pans, then the generator is plugged in and switched on. After that, the patient's hands are placed in the pans.
  The treatment is administrated by slowly increased intensity to tell the patient to feel a tingling sensation or up to 20 milliamperes and continue with this polarity for 10 minutes. After that, the polarity reversed and intensity increased again to the desired level for another 10 minutes.
  Arms: Tap water iontophoresis

SUMMARY:
the purpose of the present study is to assess the effect of laser acupoints on subjects with hyperhidrosis in comparison to tap water iontophoresis

DETAILED DESCRIPTION:
The study will be randomized control trial pre and post-experimental design. Anonymity and confidentiality of all procedures will be assured in compliance with relevant laws and institutional guidelines. All patients will sign two copies of a consent form before the beginning of data collection. Subjects will be recruited using publicly distributed posters and by online social media, subjects their hyperhidrosis examined by Hyperhidrosis Disease Severity Scale, Perceived Stress Scale. Recruited subjects will be randomly assigned to Laser Acupoint or Tap water iontophoresis groups. The participants and assessor will be blinded for the study hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* volunteer subjects from MIT physical therapy students complained from hyperhidrosis examined by Hyperhidrosis Disease Severity Scale, Perceived Stress Scale.

Exclusion Criteria:

* Subjects will be excluded if they had musculoskeletal diseases and visceral disorders or had any operations or recent injury

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Hyperhidrosis Disease Severity Scale | Change between baseline and 2 weeks of treatment measures
  The Hyperhidrosis Disease Severity Scale (HDSS) is a disease-specific, quick, and easily-understood diagnostic tool that provides a qualitative measure of the severity of the patient's condition based on how it affects daily activities. Ask the patient to select the statement above that best reflects his or her experience with sweating of the specified body area. Next to each statement is a number. A score of 3 or 4 indicates severe hyperhidrosis. A score of 1 or 2 indicates mild or moderate hyperhidrosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelshaikh University, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided